CLINICAL TRIAL: NCT04133714
Title: A Multi-center RCT Study on the Efficacy and Mechanism of Multi-channel tDCS in Rehabilitation of Cognitive Function After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-313
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2019-10

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multi-channel tDCS (Experimental): In the multi-channel tDCS stimulation group, a 1:4 (anode: cathode) approach was applied, with the central anode placed in the left dorsolateral prefrontal cortex (dlPFC) (reference 10-20 standard lead EEG), and the remaining cathode distributed around the central electrode.
  The rising time and falling time of current are 30 seconds respectively. Stimulate 30 minutes daily for 10 days (Monday to Friday, once a day, weekend off).
  Interventions: Device: multi-channel tDCS
- single-channel tDCS (Experimental): The anode electrode of the single-channel tDCS stimulation group was placed in the left dlPFC, and the cathode electrode was placed in the right orbital forehead.
  The rising time and falling time of current are 30 seconds respectively. Stimulate 30 minutes daily for 10 days (Monday to Friday, once a day, weekend off).
  Interventions: Device: single-channel tDCS
- sham stimulation (Sham Comparator): The shame stimulation group had only 30 seconds of up and down stimulation, with no intermediate stimulation.
  Interventions: Device: multi-channel tDCS; Device: single-channel tDCS

INTERVENTIONS:
Device: multi-channel tDCS — multi-channel transcranial direct current stimulation, tDCS
  Arms: multi-channel tDCS; sham stimulation
Device: single-channel tDCS — single-channel transcranial direct current stimulation
  Arms: sham stimulation; single-channel tDCS

SUMMARY:
This clinical RCT study intends to combined different forms of multi-channel tDCS with the routine cognitive training process to treat patients with post-stroke cognitive dysfunction.

The therapeutic effects among single-channel tDCS group, multi-channel tDCS and pseudo-multichannel tDCS group will be compared. Brain magnetic resonance mechanism research will also be included to reveal the possible mechanism of multi-channel tDCS technology for PSCI brain network.

Thus, the efficacy and mechanism of multi-channel tDCS in post-stroke cognitive function rehabilitation will be researched both in the clinical and basic levels.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year-old
* diagnosed cerebral apoplexy, meeting the diagnostic criteria of ICD-10
* cognitive function, perceptual function decline after stroke
* first onset and duration of 3-12 months
* right-handed
* MMSE ≤25
* MoCA ≤25
* sign informed consent voluntarily and comply with the study plan

Exclusion Criteria:

* NIHSS ≥21 points
* MoCA ≤18, or DRS-2 ≤ 124, or CES-D ≥ 16
* taking drugs that affect central nervous activity, such as nerve antagonists
* specific contraindication, such as electrode patch allergy, local skin injury or - - - - inflammation, and hyperalgesia in stimulated areas
* patients use implantable electronic devices (such as cardiac pacemakers) or have - metal implants such as stents that affect MRI examination
* patients with a previous history of epilepsy, mental illness or skull injury
* patients with dementia or obvious cognitive dysfunction before stroke
* patients with aphasia or dysarthria and cannot complete the scale evaluation
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
MMSE | Change from Baseline MMSE at 2 weeks and 3 months after intervention
  Mini-mental State Examination
MoCA | Change from Baseline MoCA at 2 weeks and 3 months after intervention
  Montreal Cognitive Assessment
AVLT | Change from Baseline AVLT at 2 weeks and 3 months after intervention
  The Auditory-Verbal Learning Test
WAIS-DST | Change from Baseline WAIS-DST at 2 weeks and 3 months after intervention
  WAIS Digit Symbol Test

SECONDARY OUTCOMES:
DEX | Change from Baseline DEX at 2 weeks and 3 months after intervention
  Dysexecutive Ques-tionnaire
GNAT | Change from Baseline GNAT at 2 weeks and 3 months after intervention
  Go/No-go Association Task

CONTACTS AND LOCATIONS:
Overall Officials: Hongjie Jiang, Dr., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University; Ruidong Cheng, Dr., Principal Investigator — Zhejiang Provincial People's Hospital; Rang Wang, Dr., Principal Investigator — Rainbowfish Rehabilitation Nursing Care; Jingming Hou, Dr., Principal Investigator — Southwest Hospital, China
Locations (4):
- China (4):
  - Rainbowfish Rehabilitation Nursing Care, Hangzhou, Zhejiang
  - SAHZhejiangU, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Southwest Hospital, Chongqing